CLINICAL TRIAL: NCT01755780
Title: The Effect of the Side of Interscalene Block on the Occurrence of Bradycardia and Hypotension During Shoulder Surgery in the Beach Chair Position
Brief Title: Effect of the Side of Interscalene Block on Bradycardia and Hypotension in Beach Chair Position
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Marina Simaioforidou, Anesthesiologist, Larissa University Hospital
Other Study IDs: Intrerscalene beach chair
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Shoulder Surgery; Beach Chair Position; Interscalene Block; Hypotension; Bradycardia; Autonomic Nervous System
MeSH Terms: conditions — Hypotension; Bradycardia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Left interscalene block: Left interscalene block on hypotension and bradycardia during beach chair positioning
  Interventions: Other: Left interscalene block
- Right interscalene block: Right interscalene block on hypotension and bradycardia during beach chair positioning
  Interventions: Other: Right interscalene block

INTERVENTIONS:
Other: Left interscalene block
  Groups: Left interscalene block
Other: Right interscalene block
  Groups: Right interscalene block

SUMMARY:
The Left interscalene block has a different effect on heart's autonomic nervous system, compared to Right interscalene block. This effect is evident on the occurrence of bradycardia and hypotension during shoulder surgery in the beach chair position

ELIGIBILITY:
Inclusion Criteria:

* elective shoulder surgery
* Age 50- 80 years old
* ASA II - IV

Exclusion Criteria:

* Coagulopathy disorders
* Infection at the puncture site for the interscalene block
* Neurological deficit on the side to be operated
* Allergy to local anesthetics
* Psychiatric disorders
* Patient's refusal
* Problems with patient communication
* Failure of the interscalene block

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for elective shoulder surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-01 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Interscalene block and beach chair positioning | Intraoperatively
  Effect of interscalene block on hypotension and bradycardia during beach chair positioning

CONTACTS AND LOCATIONS:
Overall Officials: Marina Simaioforidou, MD, Principal Investigator — Larissa University Hospital; George Vretzakis, Medicine, Study Director — Larissa University Hospital; Katerina Tsiaka, Medicine, Study Chair — Larissa University Hospital; George Basdekis, Medicine, Study Chair — Larissa University Hospital; Athanasios Drakos, Medicine, Study Chair — Larissa University Hospital
Locations (1):
- Larissa University Hospital, Larissa, Thessally, Greece